CLINICAL TRIAL: NCT01486615
Title: Premedication With Melatonin and Alprazolam Combination Versus Alprazolam or Melatonin Alone: a Randomized, Double Blind Placebo Controlled Study
Brief Title: Premedication With Melatonin and Alprazolam Combination Versus Alprazolam or Melatonin Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Krishna Pokharel, Associate Professor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2/18 (Acd. 796/067/068)
Record Dates: First submitted 2011-11-10; First posted 2011-12-06 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Anxiety
Keywords: premedication; premedicants; preoperative anxiety; melatonin; alprazolam
MeSH Terms: conditions — Anxiety Disorders | interventions — Melatonin; Azaperone; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Melatonin (Placebo Comparator): Premedication with 3 mg melatonin (Meloset) tablet orally 1-2 hour prior to anesthesia
  Interventions: Drug: meloset (melatonin)
- melatonin and alprazolam premedication (Placebo Comparator): Premedication with 3 mg melatonin and 0.5 mg alprazolam (Stresnil) tablet orally 1-2 hrs prior to anesthesia
  Interventions: Drug: stresnil ( melatonin and alprazolam)
- alprazolam premedication (Placebo Comparator): Premedication with 0.5 mg alprazolam (Alprax) tablet orally 1-2 hr prior to anesthesia
  Interventions: Drug: (alprax) alprazolam
- placebo premedication (Active Comparator): Premedication with a similar looking placebo tablet orally 1-2 hr prior to anesthesia
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: meloset (melatonin) — 3 mg melatonin tablet 1-2 hour prior surgery
  Arms: Melatonin
Drug: stresnil ( melatonin and alprazolam) — 3 mg melatonin and 0.5 mg alprazolam 1-2 hr before anesthesia
  Arms: melatonin and alprazolam premedication
Drug: (alprax) alprazolam — 0.5 mg alprazolam
  Arms: alprazolam premedication
Drug: placebo — similar looking placebo tablet
  Arms: placebo premedication

SUMMARY:
Background: Benzodiazepine, a common premedicant, suppresses endogenous melatonin levels and thus paradoxically increases episodes of arousal during sleep and thus causes restlessness and hangs over effects. Adding melatonin to it may decrease nocturnal arousal and promote the perception of sound sleep in the perioperative period.

Methods: Eighty patients (ASA 1&2) with anxiety VAS ≥ 2 posted for general anaesthesia will be randomly assigned to receive 0.5 mg alprazolam (Group A), 3 mg melatonin, a combination of 0.5 mg alprazolam and 3 mg melatonin (Group AM), or a similar looking placebo (Group P), approximately 90 minutes before surgery.

DETAILED DESCRIPTION:
Review of literature:

Benzodiazepines are among the most popular drugs used for preoperative medication to produce anxiolysis, amnesia, and sedation. However, they negatively influence sleep quality by decreasing the duration of REM sleep and slow wave sleep.

Alprazolam is more anxioselective than the more commonly used ones like midazolam, lorazepam and diazepam.Melatonin (N-acetyl-5-methoxytryptamine) is an emerging premedicant as it possesses anxiolytic and sedative properties without impairing cognitive or psychomotor skills.5 Moreover, it has an excellent safety profile.

We designed this prospective randomized double blind placebo controlled study to assess whether addition of melatonin to alprazolam has any benefit over alprazolam, melatonin or placebo alone as a premedication agent.

Rationale of the study Melatonin facilitates sleep onset and improves the quality of sleep. On the other hand, benzodiazepines suppress endogenous melatonin levels and thus paradoxically increase episodes of arousal during sleep causing restlessness and hang over effects (fatigue).

Hence, the rationale of using melatonin alprazolam combination is melatonin may decrease nocturnal arousal and promote the perception of sound sleep and thus reverse this unwanted side effect of alprazolam. Melatonin does not produce amnesia and adding a benzodiazepine to it may be desirable to achieve this desirable premedication effect.

Research design and methodology:

After getting approval from the institutional research ethics committee and written informed consent, we will study eighty patients. With the help of computer generated random numbers, patients will be assigned to one of the four groups (n=20) to receive vitamin B (Group P), 0.5 mg alprazolam (Group A), 3mg melatonin (Group M) or a combination of 0.5 mg alprazolam and 3 mg melatonin (Group AM) approximately 90 minutes before surgery. In addition to the study drugs, Groups A and AM will also receive vitamin B.

On the preanaesthetic visit one day prior to surgery, the patients will be explained about the nature of the study and the various scales to be used. A 10 cm linear Visual Analogue Scale (VAS) as well as Nepali version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS) will be used to assess their anxiety level. The extremes of the VAS anxiety scale will be marked as 'no anxiety' at the 0 end and 'anxiety as bad as ever can be' at the 10 cm end. Sedation will be assessed with a 5 point scale (0=alert, 1=arouses to voice, 2=arouses with gentle tactile stimulation, 3=arouses with vigorous tactile stimulation, 4=lack of responsiveness) and orientation, with a 3 point scale (0=none, 1=orientation in either time or place, 2=orientation in both). To test for the memory, recall of 5 different simple pictures and 2 events will be assessed. Pictures to be used will be sequentially numbered on the back and their names printed on the front.

Approximately 2 hours prior to surgery, each patient will be taken to a quiet room. Non invasive blood pressure, heart rate, respiratory rate and SpO2 will be monitored. Then picture 1 (cup on a plate) and 2 (fruits) will be shown at 10 min before and just prior to the drug administration respectively. Patients will be asked to take the study medication orally with 15 ml of plain water according to the group assignment by an investigator not involved in the patient management and data collection thereafter. Then anxiety, sedation and orientation will be assessed at 15 min, 30 min and 1 hour after the drug administration. At these time points pictures 3 (bird), 4 (hare) and 5 (car) will also be shown respectively.

In the operating room, intravenous access will be secured and pethidine 1 mg/kg administered. Then intravenous lidocaine 20 mg bolus will be administered followed by propofol with infusion pump at 100 ml per hour till responses to verbal command and eyelash reflex are lost. Vecuronium 0.1 mg/kg and isoflurane in oxygen will be administered to maintain the adequate depth of anaesthesia. After intubation, ventilation will be adjusted to maintain normocapnia. Incremental doses of pethidine and vecuronium will be administered as needed on the discretion of the investigator blinded to the patient's group assignment. No other analgesics will be administered. After completion of surgery, intravenous neostigmine 50 microgram/kg and glycopyrrolate 10 microgram/kg will be given to reverse muscle paralysis. Anaesthesia time (induction to emergence) will be noted.

In the recovery room, patients will receive the standard postoperative care; including oxygen administration via face mask 6 L/min and monitoring of heart rate, respiratory rate, non invasive blood pressure and SpO2. Modified Aldrete score and sedation score will be assessed at 10 min and 30 min after extubation. Also the occurrence of nausea, vomiting, dizziness, headache and restlessness will be recorded till 24 hours. Vomiting will be managed with ondansetron 4 mg intravenously.

The next day, the patients will be asked if they recalled the two events; being transported to operating room and intravenous cannula being inserted. They will also be asked to have a free recall of the five pictures they were shown and the score will represent the numbers of pictures they recalled. Then the first five pictures that they were shown will be mixed with next 5 new pictures (of a horse, shoe, bicycle, elephant and tiger) and they will be asked to recognize those they had already seen. The score will represent the number of pictures correctly identified. They will also be asked whether they felt that premedication drug is required to relieve anxiety and also whether they would like to receive the same premedication drug in the future.

Statistical analysis: Data will be tested for normal distribution using Kolmogorov-Smirnov test. To identify differences between groups, one-way ANOVA will be used for normally distributed continuing data and chi square tests for categorical data. If the data is found to be not normally distributed; they will be analyzed with nonparametric statistical methods. Friedman repeated measures analysis of variance followed by Wilcoxon tests with Bonferroni correction will be used for within-group comparison of values between different time points. Kruskal Wallis tests with post hoc multiple comparisons by Mann Whitney U test will be used for the comparison of values between the groups at each time points. Parametric data will be expressed as the mean±SD and nonparametric data as median (interquartile range). A p value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* (ASA 1&2),
* aging 18 to 65 years
* having anxiety VAS score of more than 2
* posted for general anaesthesia with estimated duration of < 3 hours.

Exclusion Criteria:

* patients taking analgesics, sedatives, antiepileptics or antidepressants,
* suffering from obesity (BMI ≥ 28) or neuropsychiatric disease,
* having allergy to the study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Pokharel, MD, Principal Investigator — B.P. Koirala Institute of Health Sciences; Balkrishna Bhattarai, MD, Study Director — B.P. Koirala Institute of Health Sciences
Locations (2):
- Nepal (2):
  - B. P. Koirala Institute of Health Sciences, Dharān, Koshi
  - Dr Krishna Pokharel, Dharān, Koshi

REFERENCES:
- [Background] Naguib M, Samarkandi AH, Moniem MA, Mansour Eel-D, Alshaer AA, Al-Ayyaf HA, Fadin A, Alharby SW. The effects of melatonin premedication on propofol and thiopental induction dose-response curves: a prospective, randomized, double-blind study. Anesth Analg. 2006 Dec;103(6):1448-52. doi: 10.1213/01.ane.0000244534.24216.3a. PMID 17122221
- [Background] Naguib M, Samarkandi AH. The comparative dose-response effects of melatonin and midazolam for premedication of adult patients: a double-blinded, placebo-controlled study. Anesth Analg. 2000 Aug;91(2):473-9. doi: 10.1097/00000539-200008000-00046. PMID 10910871
- [Background] Naguib M, Samarkandi AH. Premedication with melatonin: a double-blind, placebo-controlled comparison with midazolam. Br J Anaesth. 1999 Jun;82(6):875-80. doi: 10.1093/bja/82.6.875. PMID 10562782
- [Background] De Witte JL, Alegret C, Sessler DI, Cammu G. Preoperative alprazolam reduces anxiety in ambulatory surgery patients: a comparison with oral midazolam. Anesth Analg. 2002 Dec;95(6):1601-6, table of contents. doi: 10.1097/00000539-200212000-00024. PMID 12456424
- [Background] Seabra ML, Bignotto M, Pinto LR Jr, Tufik S. Randomized, double-blind clinical trial, controlled with placebo, of the toxicology of chronic melatonin treatment. J Pineal Res. 2000 Nov;29(4):193-200. doi: 10.1034/j.1600-0633.2002.290401.x. PMID 11068941
- [Background] Wade AG, Ford I, Crawford G, McMahon AD, Nir T, Laudon M, Zisapel N. Efficacy of prolonged release melatonin in insomnia patients aged 55-80 years: quality of sleep and next-day alertness outcomes. Curr Med Res Opin. 2007 Oct;23(10):2597-605. doi: 10.1185/030079907X233098. PMID 17875243
- [Background] Wurtman RJ, Zhdanova I. Improvement of sleep quality by melatonin. Lancet. 1995 Dec 2;346(8988):1491. doi: 10.1016/s0140-6736(95)92509-0. No abstract available. PMID 7491013
- [Derived] Pokharel K, Tripathi M, Gupta PK, Bhattarai B, Khatiwada S, Subedi A. Premedication with oral alprazolam and melatonin combination: a comparison with either alone--a randomized controlled factorial trial. Biomed Res Int. 2014;2014:356964. doi: 10.1155/2014/356964. Epub 2014 Jan 12. PMID 24527443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was of three months. Approximately 90 minutes prior to surgery, each patient was taken to a quiet room inside the operation theater complex.
Pre-assignment Details: One hundred and ten patients were assessed for eligibility, 98 patients had anxiety VAS ≥3. Among them, 80 patients who met the inclusion criteria, were enrolled and assigned into four groups.
Groups:
- Melatonin: Oral premedication with 3 mg melatonin tablet (Meloset) 1-2 hour prior to anesthesia
- Melatonin and Alprazolam: Oral premedication with a 3 mg melatonin and 0.5 mg alprazolam combination tablet (Stressnil) 1-2 hrs prior to anesthesia
- Alprazolam: Oral premedication with 0.5 mg alprazolam (Alprax) 1-2 hr prior to anesthesia
- Placebo: Oral premedication with a similar looking placebo tablet 1-2 hr prior to anesthesia
Period: Overall Study
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Started | 20 | 20 | 20 | 20
Completed | 20 | 19 (observed till 2 hrs after premedication, not available after 24 hours as surgery was postponed) | 18 (observed till 2 hrs after premedication, not available after 24 hours as surgery was postponed) | 18 (observed till 2 hrs after premedication, not available after 24 hours as surgery was postponed)
Not Completed | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Melatonin: premedication 1-2 hour prior to anesthesia
- Melatonin and Alprazolam: premedicated 1-2 hrs prior to anesthesia
- Alprazolam; Placebo: premedication 1-2 hr prior to anesthesia
- Total: Total of all reporting groups
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.8 (10.9) | 38.0 (13.5) | 36.9 (10.0) | 36.2 (12.9) | 36 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 16 | 15 | 61
  Male | 4 | 6 | 4 | 5 | 19
Region of Enrollment [Number; unit: participants]
  Nepal | 20 | 20 | 20 | 20 | 80
Vas baseline (cm) [Median (Inter-Quartile Range); unit: centimeters] — VAS (Visual Analogue Score) Anxiety Scale is 10 cm long and has the patient's side (front) and the clinician's side (back). The extremes of the front are colored as white and black; with a gradual darkening of color from white to black in between. The back is marked in centimeter from 0 to 10 and 0 correlates with white color (no anxiety at all) and 10 correlates to black color (anxiety as bad as ever can be). The patient is asked to point at the color on the scale according to his anxiety level. As anxiety is worsened, the score is more. The maximum value of assessment is 10 and minimum is 0.
  centimeters | 5 [4 to 6] | 5 [3.6 to 6] | 5 [4.2 to 7] | 5 [4 to 6] | 5 [4 to 6]
Anaesthesia time [Mean (Standard Deviation); unit: minutes] | 65.8 (18.1) | 77.2 (34.3) | 73.7 (21.0) | 71.7 (17.6) | 71.6 (23.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS Anxiety Score Relative to Baseline After Premedication
Description: VAS (Visual Analogue Score) Anxiety Scale is a 10 cm long scale with two sides, the patient side (front) and the clinicians side (back). The extremes of the front are colored as white and black with a gradual darkening of color from white to black. The back is marked in centimeter from 0 to 10 and 0 correlates with white color (no anxiety at all) and 10 correlates to black color (anxiety as bad as ever can be) on the front. As anxiety is worsened, the color is darker and score is more. The maximum score is 10 and minimum 0. The patient is asked to point on the scale according to his anxiety level. The anxiety score is the correlating number on the clinicians side. The more the reduction in anxiety from baseline, the better the outcome.
Time Frame: Change from baseline in VAS anxiety score at 15 minutes after premedication
Population: sample size of 16 patients in each group was determined by a power analysis (α, 0.05; β, 0.10) assuming that there will be 50% reduction in anxiety VAS from baseline in the experimental groups and 4% in the placebo group. To compensate for dropout cases and shifting from normality in data distribution, 20 cases were studied in each group.
Measure: Mean (Standard Deviation); unit: Centimeter
Groups:
- Melatonin: premedicated 1-2 hour before anesthesia
- Melatonin and Alprazolam: premedicated 1-2 hrs before anesthesia
- Alprazolam; Placebo: premedicated 1-2 hours before anesthesia
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
Centimeter | 0.35 (0.8) | 0.70 (1.6) | 0.65 (1.2) | 0.25 (0.8)

2. Secondary Outcome: Sedation Score at One Hour After Premedication
Description: Sedation level was assessed with a 5 point scale (0=alert, 1=arouses to voice, 2=arouses with gentle tactile stimulation, 3=arouses with vigorous tactile stimulation, 4=lack of responsiveness). Minimum score is 0 and Maximum is 4. The lesser the score, the better the outcome.
Time Frame: Sedation score at 1 hour after the premedication
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale | 0.5 [0 to 1] | 1 [1 to 2.75] | 1 [0 to 1.75] | 0 [0 to 1]

3. Secondary Outcome: Orientation Score
Description: Orientation was assessed with a 3 point scale (0=none, 1=orientation in either time or place, 2=orientation in both). Minimum score is 0 and maximum is 2. The lesser the score, the lesser the effect on patients cognition and the better the outcome.
Time Frame: Orientation score at one hour after premedication
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
units on a scale | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 2]

4. Secondary Outcome: Number of Patients With Intact Memory
Description: Number of patients who recalled or recognized the picture number five shown one hour after premedication. The more the number of patients with intact memory, the better the outcome.
Time Frame: 24 hour after surgery
Measure: Number; unit: Participants
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 19 | 18 | 18
Participants | 13 | 4 | 5 | 14

5. Secondary Outcome: Amount of Propofol Consumption
Description: Dose of propofol needed for loss of response to verbal command was noted at the time of induction of general anesthesia. The lesser the propofol needed for the loss of response to verbal command, the better the outcome.
Time Frame: 1 - 2 hour after premedication
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 19 | 18 | 18
mg | 79.2 (4) | 65.5 (21) | 59.0 (21) | 75.8 (25)

6. Primary Outcome: Change in VAS Anxiety Score Relative to Baseline at 30 Minutes After Premedication
Description: as for outcome 1
Time Frame: Changes from baseline in VAS anxiety score at 30 minutes after premedication
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
centimeter | 1.15 (1.4) | 1.72 (2.2) | 1.62 (1.6) | 0.82 (1.6)

7. Primary Outcome: Change in VAS Anxiety Score Relative to Baseline at One Hour After Premedication
Description: as for outcome 1
Time Frame: Changes from baseline in VAS anxiety score at one hour after premedication
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
Centimeter | 1.80 (1.7) | 2.92 (2.3) | 2.35 (2.1) | 0.85 (1.9)

8. Secondary Outcome: Number of Patients With Loss of Memory for Being Transferred to Operating Room.
Description: Patients were asked whether they recalled the event of being transferred to the operating room before anaesthesia. The lesser the number of patients with amnesia, the better the outcome.
Time Frame: 24 hour after surgery
Measure: Number; unit: Participants
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Number analyzed (Participants) | 20 | 19 | 18 | 18
Participants | 1 | 5 | 4 | 0

ADVERSE EVENTS:
Time Frame: 24 hours after premedication
Description: Incidence of nausea and vomiting were recorded.
  Vitals (Blood Pressure, Heart Rate, Respiratory rate and Temperature) were assessed every 6 hours.
Arm/Group | Melatonin | Melatonin and Alprazolam | Alprazolam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 13/20 | 12/19 | 14/18 | 16/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin (N=20) | Melatonin and Alprazolam (N=19) | Alprazolam (N=18) | Placebo (N=18)
Dizziness (Nervous system disorders) | 5 (7) | 3 (5) | 2 (4) | 4 (5)
Restlessness (General disorders) | 6 (6) | 7 (7) | 9 (9) | 8 (8)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 3 (3) | 5 (5)
Nausea and Vomiting (Gastrointestinal disorders) | 6 (8) | 7 (10) | 8 (11) | 9 (12)

LIMITATIONS AND CAVEATS:
The study was not designed to measure drug plasma concentrations. We did not perform a battery of tests to evaluate psychomotor and amnesic performances. We only did an orientation score and assessed delayed visual episodic memory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No